CLINICAL TRIAL: NCT01978301
Title: A Randomised Open Label Placebo Controlled Study to Evaluate Fractional Collagen Synthesis in Keloids and Identify Biomarkers of Keloid Biology for Potential Application in Future Clinical Trials
Brief Title: Study to Evaluate Fractional Collagen Synthesis Within Keloid Scars and Identify Biomarkers of Keloid Scars
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Temporary hold on recruitment during staff changes at the site
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 117287
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Fibrosis
Keywords: triamcinolone acetonide (TAC); heavy water; fibrosis; deuterium; collagen degradation; collagen synthesis; Keloid; patient
MeSH Terms: conditions — Fibrosis; Keloid | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triamcinolone acetonide (Active Comparator): Subjects will receive three intra-lesional injections of triamcinolone acetonide in their qualifying keloid(s), at 2-3 weeks intervals, according to their assigned treatment sequence
  Interventions: Drug: Triamcinolone acetonide
- Placebo (Placebo Comparator): Subjects will receive three intra-lesional injections of placebo in their qualifying keloid(s), at 2-3 weeks intervals, according to their assigned treatment sequence.
  Interventions: Drug: Placebo
- No treatment (No Intervention): Keloid(s) assigned 'No Treatment' will not receive any treatment.

INTERVENTIONS:
Drug: Triamcinolone acetonide — Triamcinolone acetonide will be administered as intra-lesional injection in the keloid(s).
  Arms: Triamcinolone acetonide
Drug: Placebo — Placebo will supplied as commercial injectable saline, and will be administered as intra-lesional injection in the keloid(s).
  Arms: Placebo

SUMMARY:
This is a 3-arm randomised clinical enabling study, with no investigational product. Keloid patients who are scheduled for surgical excision of one or more keloid scars (up to nine) will be recruited to the study. The aim is to investigate how collagen synthesis within keloid scars is affected by the current approved steroid treatment for keloids, triamcinolone acetonide (TAC). The primary endpoint will be fractional collagen synthesis in keloids which have received intra-lesional injections of TAC, placebo or no treatment prior to their removal. Fractional collagen synthesis will be determined using an established isotope/mass spectrometric technique which measures levels of deuterium incorporation into collagen following administration of heavy water to the subject. In addition; keloid tissue samples will be evaluated post surgery to identify further biomarkers of extracellular matrix synthesis and degradation for application in future clinical studies. Subjects will complete a screening visit and will then be randomised to receive three intra-lesional injections of TAC or placebo, or no treatment, at an interval of 2-3 weeks. Subjects will be randomised to different treatment sequences depending on the number of keloids they have scheduled for surgery, in such a way that subjects with multiple keloids will receive different arms of study treatment in their different keloids. Planned surgery for removal of their keloid(s) will be performed at week 6-8. All subjects will receive daily heavy water (Deuterium oxide) administration (twice daily or thrice daily as directed), with the first dose being taken at the Week 2 clinic visit and the final dose being taken on the day prior to surgery. A follow-up visit will be conducted at 1-4 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have at least one keloid scar scheduled for removal as part of their normal course of treatment
* Males or females aged between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Child-bearing potential with negative pregnancy test as determined by urine human chorionic gonadotropin (hCG) test at screening, AND; agrees not to become pregnant during the course of the study and for at least 1 month after completion of heavy water consumption; OR is of non child-bearing potential
* Male subjects must agree not to father a child during the study and for at least 1 month after completion of heavy water consumption.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Keloids to be randomised must not have received steroid treatment for at least two months prior to screening.
* Evidence of other skin conditions or scarring in the region of keloid scaring (including but not limited to: hypertrophic scars, eczema, psoriasis, etc.) unless the Investigator, in consultation with the GSK medical monitor, agree that the condition is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption that could preclude safe completion of the study.
* History of sensitivity to corticosteroids or history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Subjects currently receiving oral corticosteroids.
* Subjects with a recent history of tuberculosis (TB) (within last three years).
* Evidence or recent history (past two weeks) of any infection (viral, bacterial, fungal, protozoan, or helminthic).
* History of recurrent fungal infection.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
Fractional synthesis of collagen in keloid scars | Week 6-8
  Post surgical excision of keloids, tissue samples will be obtained by snap frozen biopsies. Fractional synthesis of collagen (that is, the fraction of the collagen that is newly synthesised during the labelling period) will be determined using mass spectrometry which measures the levels of deuterium incorporation into hydroxyproline or alanine in the collagen from the excised tissue samples, following administration of heavy water (Deuterium oxide) to the subject

SECONDARY OUTCOMES:
Keloid scar volume before first dose and immediately prior to surgery | Day 1 and Week 6-8
  For each keloid under evaluation, the keloid volume will be measured using three-dimensional (3D) photography
Keloid scar surface area before first dose and immediately prior to surgery | Day 1 and Week 6-8
  For each keloid under evaluation, the keloid surface area will be measured using 3D photography
Keloid scar length and height before first dose and immediately prior to surgery | Day 1 and Week 6-8
  For each keloid under evaluation, the keloid length and height will be measured using 3D photography
Keloid scar vascularity before first dose and immediately prior to surgery | Day 1 and Week 6-8
  For each keloid under evaluation, the keloid vascularity will be measured by laser Doppler

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 117287 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117287?search=study&search_terms=117287#rs